CLINICAL TRIAL: NCT01011322
Title: A Study to Investigate the Efficacy of LT-02 in Patients With Mesalazine Refractory Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lipid Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT-02-UC-01; 2008-007952-90 (Registry Identifier: EudraCT No.:)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2010-08

CONDITIONS: Ulcerative Colitis; Large Intestine; Diarrhea; Abdominal Pain
MeSH Terms: conditions — Colitis, Ulcerative; Diarrhea; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LT-02 Dose 1 (Experimental): 0.2g IMP per dose
  Interventions: Drug: LT-02
- LT-02 Dose 2 (Experimental): 0.4g IMP per dose
  Interventions: Drug: LT-02
- LT-02 Dose 3 (Experimental): 0.8g IMP per dose
  Interventions: Drug: LT-02
- Sugar pill (Placebo Comparator): placebo matching to 0g of IMP,
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LT-02 — Comparison of different dosages of drug versus placebo. 4 times daily over 12 weeks
  Arms: LT-02 Dose 1; LT-02 Dose 2; LT-02 Dose 3
Drug: placebo — placebo
  Arms: Sugar pill

SUMMARY:
The participation in this clinical study will last approximately 21 weeks with a 1 week screening period and a 12 weeks treatment duration. If the study doctor finds, that the patients disease has significantly improved he/she will enter a treatment free follow-up period of 8 weeks. In total the study consists of 5 to 6 clinical visits (V1 - V6) and 1 telephone follow-up call.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years or older who have given written Informed Consent
* Patients with proven ulcerative colitis
* Active disease course for the last 6 weeks or longer with bloody diarrhea
* Patients with an inadequate response to a treatment with mesalazine or a documented intolerance to mesalazine.

Exclusion Criteria:

* Infectious colitis, including cytomegalovirus or Clostridium difficile induced colitis,
* Crohn's disease,
* Colitis due to other reasons than ulcerative colitis like known diverticulitis, radiation colitis, ischemic colitis, microscopic colitis, or indeterminate colitis,
* Treatment with other investigational medicinal product within 3 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of IMP in mesalazine-refractory ulcerative colitis | From day 1 of treatment until end of treatment

SECONDARY OUTCOMES:
To determine the optimal dose of IMP in mesalazine-refractory ulcerative colitis | After study is completed

CONTACTS AND LOCATIONS:
Overall Officials: Max Karner, MD, Principal Investigator — University Clinic Heidelberg, Germany
Locations (26):
- Germany (16):
  - Gastroenterologische Praxis, Baden-Baden, Baden-Wurttemberg
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Gastroenterologische Praxis, Hamburg, Hamburg
  - Interdisziplinäres Crohn&Colitis Studienzentrum, Frankfurt am Main, Hesse
  - City Hospital Braunschweig, Braunschweig, Lower Saxony
  - City Hospital Lueneburg, Lüneburg, Lower Saxony
  - Gastroenterologisches Zentrum, Minden, Lower Saxony
  - Internistische Facharztpraxis, Lüdenscheid, Northrine-Westfalia
  - Internistische Gemeinschaftspraxis, Ludwigshafen, Rhineland-Platinate
  - University Clinics des Saarlandes, Homburg/Saar, Saarland
  - UK Leipzig AOR, Klinik für Gastroenterologie und Rheumatologie,, Leipzig, Saxony
  - Internistische Gemeinschaftspraxis fuer Verdauungserkrankungen, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena, Jena, Thuringa
- Lithuania (5):
  - Kaunas Medical University Hospital , Department of Endoscopy, Kaunas, Lithuania
  - Kaunas Medical University Hospital, Department of Gastroenterology, Kaunas, Lithuania
  - Klaipeda Seamen Hospital, Klaipėda, Lithuania
  - Siauliai District Hospital, Šiauliai, Lithuania
  - Santariskes Clinics Centras, Vilnius, Lithuania
- Romania (5):
  - Clinical Hospital Colentina, Bucharest, Romania
  - SC Endocenter Medicina Integrativa Bucuresti, Bucharest, Romania
  - Cabinet Medical Individual Dr. Tirnaveanu, Oradea, Romania
  - Algomed Policlinic Timisoara, Timișoara, Romania
  - Policlinica Dr. Citu, Timișoara, Romania

REFERENCES:
- [Derived] Karner M, Kocjan A, Stein J, Schreiber S, von Boyen G, Uebel P, Schmidt C, Kupcinskas L, Dina I, Zuelch F, Keilhauer G, Stremmel W. First multicenter study of modified release phosphatidylcholine "LT-02" in ulcerative colitis: a randomized, placebo-controlled trial in mesalazine-refractory courses. Am J Gastroenterol. 2014 Jul;109(7):1041-51. doi: 10.1038/ajg.2014.104. Epub 2014 May 6. PMID 24796768